CLINICAL TRIAL: NCT06638021
Title: Targeted EHR-based Communication of Diagnostic Uncertainty (TECU) in the ED: An Effectiveness Implementation Trial
Brief Title: Targeted EHR-based Communication of Diagnostic Uncertainty in the ED
Acronym: TECU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Northwestern University (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HS029791-01 (AHRQ)
Record Dates: First submitted 2024-02-07; First posted 2024-10-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Diagnostic Uncertainty
Keywords: Patient uncertainty; Symptom-based diagnosis; ED Discharge Communication; Diagnostic Uncertainty; Best practice advisory

STUDY DESIGN:
Intervention Model Description: pre-post hybrid type 1 effectiveness implementation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-TECU Implementation (No Intervention): No intervention administered.
- Post-TECU Implementation (Experimental): When an ED clinician enters an uncertain diagnosis for a patient being discharged, the TECU BPA will notify the clinician to counsel the patient about uncertainty while additionally triggering automated 1) insertion and printing of the patient handout and 2) provision of a hyperlink for the clinician-facing checklist to guide the discharge conversation.
  Interventions: Behavioral: Targeted EHR-based Communication of Diagnostic Uncertainty (TECU)

INTERVENTIONS:
Behavioral: Targeted EHR-based Communication of Diagnostic Uncertainty (TECU) — The Targeted EHR-based Communication about Uncertainty (TECU) strategy will be activated in the electronic health record (Epic) every time an ED clinician enters an uncertain diagnosis for a patient being discharged, and will notify the clinician to counsel the patient about uncertainty while additionally triggering automated 1) insertion and printing of the patient handout and 2) provision of a hyperlink for the clinician-facing checklist to guide the discharge conversation.
  Other Names: TECU
  Arms: Post-TECU Implementation

SUMMARY:
The goal of the clinical trial is to evaluate the preliminary effectiveness and the implementation feasibility of the Targeted EHR-based Communication about Uncertainty (TECU) strategy in improving the quality of care transitions from the emergency department (ED) to home. The overall specific aims related to the trial are to test the preliminary effectiveness of TECU compared to standard of care in reducing patient uncertainty and return ED visits and evaluate the adoption of TECU, exploring patient and clinician barriers and facilitators to TECU implementation.

DETAILED DESCRIPTION:
At least 37% of patients treated in the emergency department (ED) are discharged without a definitive diagnosis, thus leaving the encounter with diagnostic uncertainty. Transitions of care are high-risk periods for patient safety, especially when patients are discharged with diagnostic uncertainty, and thus are still within the diagnostic process. Effective communication between clinicians and patients is essential to improve the quality of these care transitions. In prior AHRQ-funded research, the investigators developed several tools to support high quality discharge in the setting of diagnostic uncertainty, including a communication checklist, a training program for physicians in uncertainty communication, and a patient-facing 1-page information sheet about being discharged with uncertainty.

The investigators now propose to leverage the electronic health record (EHR) to implement a multifaceted strategy to facilitate higher quality discharge transitions for patients discharged from the ED with diagnostic uncertainty. Our Targeted EHR-based Communication about Uncertainty (TECU) strategy will be activated every time an ED clinician enters an uncertain diagnosis for a patient being discharged, and will notify the clinician to counsel the patient about uncertainty while additionally triggering automated 1) insertion and printing of the patient handout and 2) an EHR-embedded link to the clinician-facing checklist to guide the discharge conversation.

The investigators will conduct a pre-post trial with a hybrid type 1 effectiveness implementation design with the goals of: 1) Testing the preliminary effectiveness of TECU compared to standard of care in reducing patient uncertainty and return ED visits and 2) Evaluating the adoption of TECU and exploring patient and clinician barriers and facilitators to TECU implementation. This project has potential to significantly impact the quality and safety of care transitions for the one-third of patients leaving the emergency department with diagnostic uncertainty.

The TJU informatics team has built a strategy within Epic to leverage the electronic health record (EHR) to implement a multifaceted strategy to facilitate safer and higher quality discharge transitions for patients discharged from the ED with diagnostic uncertainty. This strategy - the Targeted EHR-based Communication about Uncertainty (TECU) - integrates use of an Uncertainty Communication Checklist (UCC) and an Uncertainty Discharge Document (UDD) into routine Emergency Department discharge workflows. The UCC is a checklist that guides a conversational approach, to aid clinicians in addressing topics of chief concern for patients discharged with diagnostic uncertainty. The UDD is a 1-page patient-centered, health literacy appropriate discharge document that explains the concept of diagnostic uncertainty to patients. Implementing the TECU within the EHR will alert clinicians in real-time to discuss uncertainty and to standardize the routine delivery of information about uncertainty, thereby minimizing variation and reducing bias. The investigators will conduct a hybrid type 1 design with a pre-post trial of the TECU at an urban academic ED to assess preliminary efficacy of the TECU in improving patient transitions of care home from the ED and implementation of the TECU including clinician uptake as well as barriers and facilitators to implementation.

The aims of this study are to test the preliminary effectiveness of TECU compared to standard of care in reducing patient uncertainty and return ED visits, and evaluate the adoption of TECU and explore patient and clinician barriers and facilitators to TECU implementation.

ELIGIBILITY:
Patient Inclusion Criteria:

* age 18 years or older
* English language speaking
* assigned a symptom-based diagnosis in the EHR clinical impression
* planned for discharge from the ED during the enrollment visit
* able to complete follow up assessments in 2 and 30 days
* TECU best practice advisory (BPA) electronic health record alert activates during their discharge process

Patient Exclusion Criteria:

* under the age of 18 years
* non-English speaking
* clinically unstable, psychologically impaired or intoxicated, or otherwise unable to provide informed consent as judged by research staff member
* admitted to hospital
* unable to complete follow up in 2 and 30 days
* previously enrolled in this study (during a prior ED visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Uncertainty Scale (U-Scale) | enrollment
  The Uncertainty Scale (U-Scale) is a 30-item scale designed to measure patient-level uncertainty related to acute symptoms independent of underlying disease. The scale uses a 5-point Likert-style response format, asking respondents to indicate agreement with each statement from "strongly disagree" (1) to "strongly agree" (5) and leading to a nominal score range of 30-150. Higher scores indicate greater uncertainty.

SECONDARY OUTCOMES:
The Care Transition Measure (CTM)-3 | 2 days post enrollment
  The Care Transition Measure (CTM)-3 , an abbreviated form of the Care Transition Measure, will be used to assess the quality of the care transition. The CTM-3 has been highlighted as a useful measure to capture the quality of ED-to-home care transitions to aid quality improvement. Scores can range from 0-100; the score reflects the overall quality of the care transition, with lower scored indicating a poorer quality transition, and higher scores indicating a better transition.
Transitions During Uncertainty (TDU) questionnaire | 2 days post enrollment
  The TDU will be used to assess the quality of the care transition. The TDU was designed to assess care transitions upon ED discharge, to measure both the quality of existing care transition practices and the impact of care transition interventions.
Normalisation MeAsure Development questionnaire (NoMAD) | At clinician enrollment
  The NoMAD assesses staff perceptions of factors relevant to embedding the TECU intervention that change their work practices. The investigators will explore early implementation outcomes using the NoMAD with clinicians exposed to the TECU intervention.

OTHER OUTCOMES:
Return emergency department (ED) visits | 9 days post enrollment
  As the TECU is designed to improve quality of the ED discharge for patients with diagnostic uncertainty, the investigators hypothesize that ED recidivism will decrease for patients receiving the TECU-guided discharge. The investigators will evaluate rates of ED return at 9 days and 30 days. Rates of ED return and subsequent outpatient care encounters will be assessed through patient self-report at T2 (30 days) and EHR review.
Return emergency department (ED) visits | 30 days post enrollment
  As the TECU is designed to improve quality of the ED discharge for patients with diagnostic uncertainty, the investigators hypothesize that ED recidivism will decrease for patients receiving the TECU-guided discharge. The investigators will evaluate rates of ED return at 9 days and 30 days. Rates of ED return and subsequent outpatient care encounters will be assessed through patient self-report at T2 (30 days) and EHR review.
Composite healthcare utilization | 30 days post enrollment
  The investigators acknowledge that it is possible that, when better informed about their lack of a diagnosis, total healthcare utilization may increase as patients continue to pursue a diagnosis through outpatient visits with their primary physician or specialists. The investigators will assess 30-day composite counts of all healthcare interactions including: ED and clinic visits, admissions, testing appointments, telephone or EHR-message interactions. Data will be obtained through patient self report as well as EHR queries.
Spielberger State-Trait Anxiety Inventory (STAI-AD) | enrollment
  The 6-item short-form of the Spielberger State-Trait Anxiety Inventory (STAI-AD) scale of this gold-standard measure provides a reliable and sensitive measure of anxiety in relation to an event. The 6-item STAI-ID is scored using a 4-point Likert scale (1: Not at all, 2: Somewhat, 3: Moderately so, 4: Very much so), with higher scores indicating more anxiety. Scores can range from 6-24; Scores above 15 indicate the presence of anxiety symptoms.
Spielberger State-Trait Anxiety Inventory (STAI-AD) | 2 days post enrollment
  The 6-item short-form of the Spielberger State-Trait Anxiety Inventory (STAI-AD) scale of this gold-standard measure provides a reliable and sensitive measure of anxiety in relation to an event. The 6-item STAI-ID is scored using a 4-point Likert scale (1: Not at all, 2: Somewhat, 3: Moderately so, 4: Very much so), with higher scores indicating more anxiety. Scores can range from 6-24; Scores above 15 indicate the presence of anxiety symptoms.
Spielberger State-Trait Anxiety Inventory (STAI-AD) | 30 days post enrollment
  The 6-item short-form of the Spielberger State-Trait Anxiety Inventory (STAI-AD) scale of this gold-standard measure provides a reliable and sensitive measure of anxiety in relation to an event. The 6-item STAI-ID is scored using a 4-point Likert scale (1: Not at all, 2: Somewhat, 3: Moderately so, 4: Very much so), with higher scores indicating more anxiety. Scores can range from 6-24; Scores above 15 indicate the presence of anxiety symptoms.
Care Transition Measure | 30 days post enrollment
  The Care Transition Measure (CTM)-3 , an abbreviated form of the Care Transition Measure, will be used to assess the quality of the care transition. The CTM-3 has been highlighted as a useful measure to capture the quality of ED-to-home care transitions to aid quality improvement. Scores can range from 0-100; the score reflects the overall quality of the care transition, with lower scored indicating a poorer quality transition, and higher scores indicating a better transition.
Uncertainty Scale (U-Scale) | 30 days post enrollment
  The Uncertainty Scale (U-Scale) is a 30-item scale designed to measure patient-level uncertainty related to acute symptoms independent of underlying disease. The scale uses a 5-point Likert-style response format, asking respondents to indicate agreement with each statement from "strongly disagree" (1) to "strongly agree" (5) and leading to a nominal score range of 30-150. Higher scores indicate greater uncertainty.
Uncertainty Scale (U-Scale) | 2 days post enrollment
  The Uncertainty Scale (U-Scale) is a 30-item scale designed to measure patient-level uncertainty related to acute symptoms independent of underlying disease. The scale uses a 5-point Likert-style response format, asking respondents to indicate agreement with each statement from "strongly disagree" (1) to "strongly agree" (5) and leading to a nominal score range of 30-150. Higher scores indicate greater uncertainty.
Uncertainty Scale (U-Scale) Treatment Quality subdomain | 2 days post enrollment
  The Uncertainty Scale (U-Scale) assesses patient-level uncertainty related to acute symptoms - while the U-Scale in its entirety is being assessed, the investigators also will assess for differences specifically in the uncertainty related to treatment quality subdomain, as this has been associated with return ED visits and contains the questions most immediately linked to the care and communication received during the ED visit.
Uncertainty Scale (U-Scale) Treatment Quality subdomain | 30 days post enrollment
  The Uncertainty Scale (U-Scale) assesses patient-level uncertainty related to acute symptoms - while the U-Scale in its entirety is being assessed, the investigators also will assess for differences specifically in the uncertainty related to treatment quality subdomain, as this has been associated with return ED visits and contains the questions most immediately linked to the care and communication received during the ED visit.
User feedback | 30 days (patients), enrollment (clinicians)
  Patient and clinician experience data obtained via interviews and focus groups
Clinical Sustainability Assessment Tool (CSAT) | At clinician enrollment
  The Clinical Sustainability Assessment Tool (CSAT) assesses organizational capacity for sustainability. The investigators will use the CSAT to conduct summative implementation assessment with clinicians exposed to the TECU intervention. The CSAT total score ranges from 1 to 7, with higher scores indicating a greater capacity for clinical sustainability.
Uncertainty Scale (U-Scale) Treatment Quality subdomain | enrollment
  The Uncertainty Scale (U-Scale) assesses patient-level uncertainty related to acute symptoms - while the U-Scale in its entirety is being assessed, the investigators also will assess for differences specifically in the uncertainty related to treatment quality subdomain, as this has been associated with return ED visits and contains the questions most immediately linked to the care and communication received during the ED visit.
Transitions During Uncertainty (TDU) questionnaire | enrollment
  The TDU will be used to assess the quality of the care transition. The TDU was designed to assess care transitions upon ED discharge, to measure both the quality of existing care transition practices and the impact of care transition interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Rising, MD, MS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCarthy DM, Malone S, Papanagnou D, Leiby BE, Doty AMB, Watts P, Yadav R, Pugliese JK, Woodworth J, Camacho TE, Kean E, Rising KL. Targeted EHR-based communication of diagnostic uncertainty (TECU) in the emergency department: Protocol for an effectiveness implementation trial. Contemp Clin Trials. 2025 Jun;153:107910. doi: 10.1016/j.cct.2025.107910. Epub 2025 Apr 7. PMID 40204252